CLINICAL TRIAL: NCT01686412
Title: Determination of Autonomic Responses to Exposure to Electromagnetic Fields With Low Energy Modulated Frequency in Patients With Breast and Advanced Hepatocellular Cancer.
Brief Title: Determination of Autonomic Responses to Exposure to Electromagnetic Fields With Low Energy Modulated Frequency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Principal Investigator, Frederico Perego Costa, Attending physician, Hospital Sirio-Libanes
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HSL 2012/10
Record Dates: First submitted 2012-07-12; First posted 2012-09-18 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-06

CONDITIONS: Hepatocellular Carcinoma; Breast Cancer
Keywords: Breast Cancer; Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy patients (Active Comparator)
  Interventions: Device: Electromagnetic Fields of Low Energy (EEFLE)
- Oncology patients (Active Comparator)
  Interventions: Device: Electromagnetic Fields of Low Energy (EEFLE)

INTERVENTIONS:
Device: Electromagnetic Fields of Low Energy (EEFLE) — Are employed three sets of programs of different frequencies are modulated specifically for each group of patients in accordance with diagnostic (hepatocellular carcinoma, breast carcinoma and healthy subjects). These frequencies ranging between 0.1 and 114.000Hz.

SUMMARY:
This is an exploratory study, national, unicentric, double-blind, to be conducted at the Institute for Teaching and Research of the Hospital Sírio-Libanês in order to detect possible autonomic responses resulting from Exposure to Electromagnetic Fields of Low Energy (EEFLE) in healthy subjects and in patients with advanced hepatocellular carcinoma or in patients with advanced breast carcinoma. Autonomic responses have been described in patients with cancer during the exposure of EEFLE. This autonomic response, or biofeedback, due to exposure to EEFLE seems to be associated with a specific set of modulation frequencies when applied to patients with malignancies. Moreover, healthy individuals exposed to modulated EEFLE a specific set of frequency do not appear to autonomic response. Biofeedback is defined by a change in amplitude of the radial pulse during exposure to EEFLE, modulated according to a set of specific frequencies. This phenomenon is not yet fully elucidated. In exploratory survey of one patient was observed a change of the pressure pulse immediately after the start of and during exposure to EEFLE, modulated according to a set of specific frequencies recorded by digital photoplethysmography. This study aims to evaluate an autonomic response in individuals exposed in a single moment, by electromagnetic fields. This study does not intend to study a diagnostic or therapeutic procedure. For this reason, evolutive clinical data will not be considered during and after the study.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

* Should be considered healthy, with no known relevant comorbidity.
* Patients should not be suffering from active malignancy or history of malignancy in the past.
* Must be over 18 years.
* Must have ability to understand and provide a written informed consent.

Patients with hepatocellular carcinoma:

* Patients must be diagnosed with inoperable HCC.
* Presence of primary tumor or metastatic at the time of the procedure.
* Patients with liver cirrhosis should be restricted to Child-Pugh A or B.
* Patients with AFP> 400ng/ml and image feature does not require histopathological confirmation. However, in patients with active serology B virus, this value must be greater than AFP 4000 ng / ml. The remaining patients should have histological confirmation of HCC.
* Patients may be under observation or treatment in the presence of systemic or intra-hepatic.
* Must have ability to understand and provide a written informed consent.

Patients with Ductal Carcinoma Breast

* Patients must have a diagnosis of breast ductal carcinoma inoperable.
* The presence of the primary tumor or metastatic during the procedure.
* Patients may be under observation or in the presence of systemic or hormonal treatment only.
* Must have ability to understand to provide a written informed consent.

Exclusion Criteria:

* Can not stop antihypertensive medications or beta-blockers for at least 48 hours or being in possession of a pacemaker or other implantable device.
* Pregnant or lactating women.
* Smaller than 18 years.
* Patients undergoing radiotherapy treatment or up to 2 weeks of discontinuation.
* Inability to understand and provide written informed consent.
* Liver cirrhosis Child Pugh C.
* Patients without a definite diagnosis.
* Absence of the primary tumor or metastatic during the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Autonomic response monitoring (blood pressure digital and manual monitoring) | 60 minutes

SECONDARY OUTCOMES:
Cardiovascular electronic monitoring (digital photoplethysmography and electrocardiography) | 60 minutes
Baroreflex sensitivity (by the method of sequence) | 60 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sírio-Libanês, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Capareli F, Costa F, Tuszynski JA, Sousa MC, Setogute YC, Lima PD, Carvalho L, Santos E, Gumz BP, Sabbaga J, de Castria TB, Jardim DL, Freitas D, Horvat N, Bezerra ROF, Testagrossa L, Costa T, Zanesco T, Iemma AF, Abou-Alfa GK. Low-energy amplitude-modulated electromagnetic field exposure: Feasibility study in patients with hepatocellular carcinoma. Cancer Med. 2023 Jun;12(11):12402-12412. doi: 10.1002/cam4.5944. Epub 2023 May 15. PMID 37184216